CLINICAL TRIAL: NCT03575936
Title: Enhanced Pharmacist-Managed Anticoagulation Service in a University-based Family Medicine Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Anticoagulation
Record Dates: First submitted 2018-05-23; First posted 2018-07-03 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2018-05

CONDITIONS: Anticoagulation; Home INR Monitoring
Keywords: Pharmacists Intervention
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care Group (Active Comparator): Standard of Care arm. Pharmacist intervention in clinic
  Interventions: Procedure: Standard of Care
- Home Monitoring Group (Experimental): Pharmacist intervention with home INR monitoring
  Interventions: Device: Home INR Monitoring

INTERVENTIONS:
Device: Home INR Monitoring — The self-monitoring group will monitor INR at home using the AlereTM Home Monitoring Service. They will call in the weekly results to Alere or submit online via the patient portal, which is the standard protocol among home monitoring patients. Alere will then upload the information to a password-protected HIPAA compliant website that only study investigators will be able to access. Pharmacists will have real-time access to the test results via the web interface. Pharmacists can follow up in real time if the patient forgets to self-test. An alert will also be sent to the pharmacists via email to follow up on any out of range results. This will help streamline pharmacists' workload to dedicate face-to-face time for patients that require such intervention. All home monitoring patients will be seen in clinic by the pharmacist at the end of the 3-month randomization period in order to assess compliance with meter-use and re-evaluate meter-use competency.
  Other Names: Alere Home INR Machine
  Arms: Home Monitoring Group
Procedure: Standard of Care — The patients in the standard of care group will have a clinic visit with the pharmacist at least once every 4 weeks or earlier, as deemed necessary by the pharmacist. The duration of the randomization period will be three months. At the end of the 3-month randomization period, patients will be provided the opportunity to cross over from the home INR monitoring group to the pharmacist-managed clinic group, or vice versa. The remainder of the study duration (post-3 month analysis) will purely be for observational purposes, in order to account for the loss of randomization and potential bias. The total duration of the study will be one year.
  Arms: Standard of Care Group

SUMMARY:
Introduction:

The ambulatory care pharmacist service is a vision that is supported by several national pharmacy associations and expected by many clinical environments. However, pharmacists practicing in such settings often lack the data to demonstrate their value for the services they provide. Consequently, clinical services provided by pharmacists are not viewed as a billable expense and reimbursements are bundled with drug dispensing. Thus, if a pharmacy service is to sustain for the long-term, it is imperative to develop a value model to support monetary compensation for the cognitive services provided.

Background and Significance:

Anticoagulation with warfarin is a high risk therapy involving complex dosing, monitoring, and ensuring adherence to outpatient therapy. Monitoring anticoagulation intensity utilizing the prothrombin time (PT) and the international normalized ratio (INR) is used to determine the effectiveness of anticoagulation therapy. The proportion of time the INR is within the therapeutic range (TTR) is considered a surrogate measure of anticoagulation control and is associated with lower rates of major bleeds and thromboembolism.

Pharmacist managed anticoagulation clinics eliminate the waiting period between lab work from an external facility and decisions from physicians. Pharmacists practicing in anticoagulation clinics with point-of-care INR testing usually practice under a collaborative agreement, which allows them to adjust and reverse warfarin dosing based on established protocols. This reduces the wait time and is expected to increase patient satisfaction. Despite the wide acceptance of pharmacist-managed anticoagulation clinics, there is inconsistent evidence to support prevention of major bleeding.

Methods:

This is an IRB-approved prospective, unblinded randomized controlled trial of the clinical impact of home anticoagulation monitoring. The study will enroll all patients (who meet eligibility criteria) who require long-term anticoagulation therapy from a pharmacist-managed anticoagulation clinic.

Expected Outcomes:

The purpose of this study is to evaluate if self- monitoring in addition to pharmacist review will increase the TTR. This will allow university- based pharmacists to provide care for more patients effectively in addition to their academic duties.

ELIGIBILITY:
Inclusion Criteria:

* Established patients within the USF Morsani Center Family Medicine department
* Adults over the age of 18 years
* Long-term (> 12 months) warfarin therapy
* Taking warfarin for at least 90 days prior to enrollment
* Willing and able to perform home INR monitoring with correct technique (or caregiver)

Exclusion Criteria:

* Failure by either the patient or caregiver to demonstrate successful INR monitoring technique
* Issues with mental and/or physical dexterity as evaluated and determined by the pharmacist
* Unwillingness to take full financial responsibility for costs not covered (by patient's insurance and/or grant money) incurred with home INR monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
INR | 12 months
  INR obtained weekly via home monitoring arm. INR obtained every 4 weeks or sooner for patients seen in clinic. Two arms compared to determine time within therapeutic range.

SECONDARY OUTCOMES:
Patient Satisfaction and Quality of Life with Anticoagulation utilizing the Duke Anticoagulation Satisfaction Scale (DASS) | 12 months
  Patients were given the DASS survey at baseline, 3 mo (end of randomization) & end of study (12 mo), in order to assess satisfaction with warfarin therapy & management. The DASS is a validated survey, including 25 items, each containing 7 response categories: "not at all, a little, somewhat, moderately, quite a bit, a lot, & very much". Questions are arranged to correspond to 3 possible dimensions pertaining to anticoagulation: limitations, hassles & burdens, & positive psychological impacts. The DASS is able to summarize satisfaction with anticoagulation & identify aspects that may hinder individual patients from maintaining an INR within therapeutic range. Many interventions can potentially be designed to improve anticoagulation quality of care, & thus reduce the time spent outside of therapeutic range, & ultimately thromboembolic & bleeding events by identifying the limitations, hassles & burdens, as well as positive psychological impacts experienced by patients.

IPD SHARING:
Plan to Share IPD: No